CLINICAL TRIAL: NCT06623838
Title: An Evolutionarily Informed Conceptualization of Personality Pathology: A Cross-cultural Acceptability and Reliability Study
Brief Title: An Evolutionarily Informed Conceptualization of Personality Pathology
Acronym: EIC-PP
Status: Recruiting | Type: Observational
Sponsor: Tages Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: EIC-PP
Record Dates: First submitted 2024-09-17; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Personality Disorder
Keywords: evolutionary systems therapy; personality disoders; personality pathology; evolutionary psychopathology; psychotherapy; case conceptualization
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Spanish group: Group/Cohort Description: 22 students in MA in clinical psychology performing the evolutionarily informed case conceptualization.
  Interventions: Diagnostic Test: Evolutionarily informed case conceptualization
- Polish group: Group/Cohort Description: 22 students in MA in clinical psychology performing the evolutionarily informed case conceptualization.
  Interventions: Diagnostic Test: Evolutionarily informed case conceptualization
- Chinese group: Group/Cohort Description: 22 students in MA in clinical psychology performing the evolutionarily informed case conceptualization.
  Interventions: Diagnostic Test: Evolutionarily informed case conceptualization
- Italian group: Group/Cohort Description: 22 students in MA in clinical psychology performing the evolutionarily informed case conceptualization.
  Interventions: Diagnostic Test: Evolutionarily informed case conceptualization
- American group: Group/Cohort Description: 22 students in MA in clinical psychology performing the evolutionarily informed case conceptualization.
  Interventions: Diagnostic Test: Evolutionarily informed case conceptualization

INTERVENTIONS:
Diagnostic Test: Evolutionarily informed case conceptualization — Case conceptualization of personality functioning of a few transcripts of initial sessions and report of psychometric measures of patients diagnosed with personality disorder.

SUMMARY:
The purpose of this study is to explore the reliability of a new evolutionarily-informed model for conceptualizing personality pathology. In a preliminary phase prior to the present study we investigated reliability by comparing how therapist pairs conceptualized and assessed the same patient and how therapists and patients assessed the acceptability of the model.

In this new study we want to confirm that the validity data initially collected are valid across cultures and nations.

Therefore, psychology students (n=110) from 5 countries (China, Italy, Poland, Spain, United States) will participate in a specific training on the model and then apply the model on transcripts of the first two sessions and on assessment reports and two supervisors will evaluate the inter-rater reliability and acceptability in using the model on the same patients.

DETAILED DESCRIPTION:
The study aims to investigate the cross-cultural validity of a model of assessment and conceptualization of personality disorders. Given the importance of cultural, social and health conditions in the development and maintenance of these disorders, the model will be tested in 5 different countries. This study follows two previous researches that preliminarily explored the feasibility and reliability of the model in couples of Italian patients and therapists (a detailed description of the previous studies is available in the IPD). Below is a brief description of the project registered here:

* Sample (n=110): China (n=22), Italy (n=22), Poland (n=22), Spain (n=22), United States (n=22).
* Primary goal: Interview to assess perceived utility of conceptualization in the whole samples, and then comparing different cultural backgrounds to assess cross-cultural reliability.
* Secondary goals: Scoring in adherence of students by supervisors (same scoring system as in Research 1) to compare Intra Class Correlation within and between national sub-groups.
* Procedure: All participants will access specific online sessions, one for each country sub-group. The first session will correspond to access to a presentation of the theoretical background of the conceptualization model (1 hour in recorded format that participants can access independently). The second session will correspond to an experiential training in which the model will be presented in detail with various clinical cases and a first exercise on the use of this model will be conducted (2.5 hours in live format with all participants simultaneously). The third session will instead be aimed at applying the model on a case that will be presented to all participants and will correspond to a transcript of the two initial sessions and a report on the results of the questionnaires (0.5 hour in live format that participants can access independently). The fourth session will be accessed by some participants (n= 5 per country) and will correspond to a structured interview conducted by a researcher on the acceptability and usefulness of the model (live format that participants can access independently).

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students in their final year
* Recently graduated students.

Exclusion Criteria:

* having left the university program during the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Undergraduate students in psychology
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Cross-cultural inter-rater reliabilitt | From the enrollment to the end of the end of the diagnostic procedure that last 1 hours and will be performed within 1 month from the recruitment.
  Inter-rater reliability of adherence to the case conceptualization within any single group will be compared with the Italian group where the diagnostic procedure was initially validated to confirm that there are no differences in reliability between Italian group and the other groups. Inter-rater reliability will be scored as kappa values and intraclass correlation coefficients.

CONTACTS AND LOCATIONS:
Locations (1):
- Tages Onlus, Florence, Italy

IPD SHARING:
Plan to Share IPD: Yes
Description of research, statistical plan and dataset will be published on OSF. Description of research and statistical plan are available, whereas dataset at the end of the data collection (between January and March, 2025).
  To access OSF files: https://osf.io/hnyz6/
Supporting Information: Study Protocol, SAP
Time Frame: Description of research, statistical plan and dataset will be published on OSF. Description of research and statistical plan are available, whereas dataset at the end of the data collection (between January and March, 2025).
Access Criteria: Open access
URL: https://doi.org/10.17605/OSF.IO/HNYZ6

REFERENCES:
- [Result] Cheli S, Cavalletti V, Lysaker PH, Dimaggio G, Petrocchi N, Chiarello F, Enzo C, Velicogna F, Mancini F, Goldzweig G. A pilot randomized controlled trial comparing a novel compassion and metacognition approach for schizotypal personality disorder with a combination of cognitive therapy and psychopharmacological treatment. BMC Psychiatry. 2023 Feb 20;23(1):113. doi: 10.1186/s12888-023-04610-5. PMID 36803673
- [Result] Cheli S, Goldzweig G, Chiarello F, Cavalletti V. Evolutionary systems therapy for paranoid personality disorder: A seven cases series. Bull Menninger Clin. 2024 Winter;88(1):61-80. doi: 10.1521/bumc.2024.88.1.61. PMID 38527104
- Available data/document: Study Protocol: HNYZ6 — https://doi.org/10.17605/OSF.IO/HNYZ6